CLINICAL TRIAL: NCT06105736
Title: Regulating Together in Tuberous Sclerosis Complex: A Pilot Feasibility Study in Children and Adolescents With TSC-Associated Neuropsychiatric Disorder (TAND)
Brief Title: Regulating Together in Tuberous Sclerosis Complex
Acronym: RT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Rochester (Other)
Responsible Party: Principal Investigator, Jamie Capal, Pediatric Neurologist-Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-0274; HT9425-23-1-0344 (Other Grant/Funding Number: U.S. Department of Defense); CDMRP-TS220041 (Other: U.S. Department of Defense)
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: TSC; Behavioral Symptoms
MeSH Terms: conditions — Behavioral Symptoms | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parents (Experimental): In this 22-week almost completely remote study, following a 5-week control phase, parents will receive intensive treatment twice per week for 5 weeks followed by a one-time, 1-on-1 counseling session with an RT psychologist (week 11). Then, parents will use skill practice and application in the home environment for 10 weeks. Following this, a final interview is conducted (week 22).
  Interventions: Behavioral: Behavioral Intervention in a small group platform
- Children (Experimental): In this 22-week almost completely remote study, following a 5-week control phase, children will receive intensive group treatment, twice a week for 5 weeks delivered remotely. During the children's sessions, they will use child structured videos, the PlayPosit curriculum and learning rewards. The following assessments will be completed by the parents, regarding their children, at each phase; EDI, ABC-2, FS, BRIEF-2, CRS, PSI-4SF and CGI-I. Following the completion of group treatment, there will be a one-time, 1-on-1 counseling session with an RT psychologist.
  Interventions: Behavioral: Behavioral Intervention in a small group platform

INTERVENTIONS:
Behavioral: Behavioral Intervention in a small group platform — RT is small-group-based, intensive behavioral intervention session delivered twice weekly over a secure remote platform for 60-minutes over 5 weeks. Each session is led by a psychologist trained and certified in RT. Caregiver groups meet at the same frequency and duration but at different times. Each session has a specific focus for teaching participants to identify emotions and incorporation of cognitive behavioral therapy (CBT) and mindfulness skills that are reinforced through repeated practice. Each session will include a review, relaxation, new material didactic, activities to reinforce material, mindfulness, and homework.

SUMMARY:
The purpose of this study is to use a program called Regulating Together (RT), a remote, non-pharmacologic intervention to treat symptoms of emotion dysregulation in children and adolescents with Tuberous Sclerosis Complex (TSC) and TSC-Associated Neuropsychiatric Disorder (TAND).

DETAILED DESCRIPTION:
This is a non-pharmacological intervention that will utilize small group-based therapy with participants, followed by a separate caregiver session. The clinical trial will consist of four phases; 1) single in person screening/baseline visit; 2) RT control phase which is a 5-week observational period (Week 1-5); 3) RT intensive phase which is a remote group treatment intervention twice per week over 5 weeks (Week 6-10); 4) RT individualization phase, which is an individualized consultation with the participant and caregiver (Week 11); and 5) the RT generalization phase which is a 10 week follow up period consisting of utilizing the learned skills at home. At the end of the 10-week generalization phase, a semi-structured interview for thematic analysis will occur at the end of the study to capture facilitators and barriers to the intervention (Week 12-22).

ELIGIBILITY:
Inclusion Criteria:

* Children ages 8-17 years inclusive with a documented clinical and/or genetic diagnosis of TSC and exhibiting symptoms of behavioral dysregulation (identified on the TAND Checklist having temper tantrums, aggressive outbursts, self-injury, and/or impulsivity) are eligible for inclusion.

Additional inclusion/eligibility criteria include:

* Participants and their caregivers have access to a computer, phone, or tablet with video capability and stable internet connection. If lack of a device or internet service is the sole barrier to eligibility/participation, interested individuals will be connected to a TSC Clinic social worker to link them to existing government and charity programs specifically addressing this disparity in underserved communities and households in need (e.g., the Affordable Connectivity Program).
* Participants must also be willing to participate in treatment sessions and have minimal levels of functional verbal communication (child and their caregiver must be fluent in English
* Child must have a minimum IQ>65 on the WASI-II at the screening/baseline visit).

Exclusion Criteria:

* Participants be on a stable medication regimen at least 4 weeks prior to enrollment
* Do not have a plan to start a new psychosocial intervention (e.g., individual psychotherapy, family psychotherapy, group psychotherapy or social skills training) or behavior medication within 30 days prior to enrollment or at any point during the study. ----Participants with significant disruptive, aggressive, self-injurious or sexually inappropriate behaviors deemed potentially dangerous or overly disruptive to the group dynamic/session, having significant co-occurring neuropsychiatric illness warranting other treatment approaches as determined by study clinician (e.g., substance use disorders, psychotic disorders, schizophrenia), or having significant sensory impairment that would limit participation in intervention curriculum/materials (e.g., blindness or uncorrected hearing loss) also will be excluded.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Prevalence of ED in TSC Cohort | Baseline
  Prevalence of emotion dysregulation is highly prevalent in TSC patients who exhibit problematic behaviors. The EDI-R score at the screening study visit will determine the EDI-R and determine the presence or absence of emotion dysregulation in the cohort.
Change in EDI-R Score from Control Phase to RT Intensive and RT Generalization Phases Combined | Intensive Phase (Week 6-10) and Generalization Phase (Week 12-22)
  EDI-R score will be compared from pre-treatment (control phase) to post-treatment (RT Intensive Phase and RT Generalization Phases combined). EDI-R is a caregiver administered, emotion dysregulation inventory with construct, range, and directionality that includes questions that the rater is asked to answer based on behaviors that are observed to cause problems. These questions include, but are not limited to, creating a dangerous situation, interference with daily activities, increasing the stress of those around the individual, and hurting relationships. There are 13 questions on the EDI-R; they are rated at, not at all, mild, moderate, severe, and very severe.
Change in CP-CTI score from pre-treatment to post-treatment | Administered after completion of RT (Week 22)
  The primary endpoint will be CP-CTI responses from caregivers upon completion of RT Generalization Phase using a thematic analysis. This will identify obstacles to treatment access. Scores will be compared pre-treatment to post-treatment. CP-CTI is a staff administered, caregiver perspective clinical trial interview. This will occur through a telephone call from the study team to the caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Capal, MD, Principal Investigator — University of North Carollina at Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina Chapel Hill-Carolina Institute for Developmental Disabilities, Carrboro, North Carolina
  - Cincinnati Children's Hospital Medical Center (CCHMC), Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: SAP
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Result] Shaffer RC, Schmitt LM, Reisinger DL, Coffman M, Horn P, Goodwin MS, Mazefsky C, Randall S, Erickson C. Regulating Together: Emotion Dysregulation Group Treatment for ASD Youth and Their Caregivers. J Autism Dev Disord. 2023 May;53(5):1942-1962. doi: 10.1007/s10803-022-05461-x. Epub 2022 Feb 9. PMID 35141815
- [Result] Shaffer RC, Wink LK, Ruberg J, Pittenger A, Adams R, Sorter M, Manning P, Erickson CA. Emotion Regulation Intensive Outpatient Programming: Development, Feasibility, and Acceptability. J Autism Dev Disord. 2019 Feb;49(2):495-508. doi: 10.1007/s10803-018-3727-2. PMID 30143951